CLINICAL TRIAL: NCT07304804
Title: The Effect of Baby Massage Training Provided to Midwifery Students on Their Knowledge of Baby Massage: A Randomized Controlled Trial
Brief Title: Effect of Baby Massage Training on Knowledge Levels of Midwifery Students
Acronym: BaMaMiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zülbiye demir barbak, Lecturer Dr., Department of Midwifery, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AtaU-HEM-ZDB-05
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Infant Massage Education; Midwifery Students
Keywords: Baby massage; Midwifery education; Knowledge level; Randomized controlled trial; Infant care; Simulation-based training

STUDY DESIGN:
Intervention Model Description: Participants were stratified by class year and randomly assigned to either the intervention group (baby massage training) or control group (no training). The study followed a parallel design with pre-test and post-test evaluation.
Masking Description: This study was open-label. Neither participants nor researchers were blinded to group assignments, as the educational intervention required active participation and observation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby Massage Training (Experimental): Participants in this group received baby massage training, which included three 30-45 minute sessions consisting of a baby massage video, mannequin-based demonstration, and guided practice. The sessions aimed to improve students' knowledge and understanding of baby massage techniques.
  Interventions: Behavioral: Baby Massage Training
- Control: No Training (No Intervention): Participants in this group did not receive any baby massage training. They completed the same pre-test and post-test assessments as the experimental group to evaluate changes in knowledge levels without exposure to the intervention.

INTERVENTIONS:
Behavioral: Baby Massage Training — A structured educational intervention consisting of three sessions (30-45 minutes each). The training included video presentation, mannequin demonstration, and guided practice on baby massage techniques.
  Other Names: Baby Massage Education
  Arms: Baby Massage Training

SUMMARY:
The goal of this clinical trial was to learn whether baby massage training could improve midwifery students' knowledge about baby massage. The study focused on students in their third and fourth years who had already completed child health and neonatal care courses.

The main question was whether students who received baby massage training would have higher knowledge scores after the training compared with students who did not receive the training.

Researchers randomly assigned 64 midwifery students into two groups:

Training group (32 students): received structured baby massage education that included a video demonstration, mannequin practice, and guided feedback.

Control group (32 students): did not receive any baby massage training during the study period.

Each student completed a questionnaire about baby massage before and after the training. The questionnaire contained 15 yes/no questions about preparation, application, and post-application steps of infant massage.

Training sessions lasted 30 to 45 minutes and were delivered by an experienced instructor in a classroom environment. The intervention took place in April-May 2024 at Atatürk University, Faculty of Health Sciences, in Türkiye.

After the training, students in the training group had significantly higher knowledge scores than those in the control group. The results showed that structured baby massage education increased the students' knowledge and awareness of infant massage practices.

DETAILED DESCRIPTION:
Detailed Description

Background and Rationale Touch is one of the earliest senses to develop and supports bonding, regulation, and growth in infants. Infant massage is a touch-based caregiving practice commonly taught by midwives and nurses. Although its benefits for infants and parents are well described, there is limited evidence on structured infant-massage education for midwifery undergraduates. This study was designed to test whether a brief, structured baby massage training improves midwifery students' knowledge about preparation, safe application, and post-application steps of infant massage.

Objectives Primary objective: To determine the effect of a structured baby massage training program on midwifery students' infant-massage knowledge measured immediately after training.

Hypothesis: Students receiving the training will have higher post-test knowledge scores than students who do not receive the training.

Study Design Randomized, parallel-group, educational intervention trial with a 1:1 allocation ratio. Stratified randomization by class year (3rd vs 4th year) using a random-number table. Open-label; outcome assessors scored written forms and checklist responses.

Setting and Dates Department of Midwifery, Faculty of Health Sciences, Atatürk University (Erzurum, Türkiye). Recruitment and delivery occurred April-May 2024 in a classroom equipped with suitable light, seating, and privacy.

Participants Target population: undergraduate midwifery students who had completed Child Health and Neonatal courses.

Inclusion criteria: 3rd or 4th year midwifery student; completed relevant courses; literate in Turkish; provided informed consent.

Exclusion criteria: withdrawal during training; missing pre- or post-test data.

Sample Size and Power A priori power analysis (medium effect size d=0.50, 95% confidence, 80% power) indicated ≥27 participants per arm. Allowing for attrition, 32 per arm were enrolled (total N=64).

Recruitment and Allocation

An invitation and study information were delivered via WhatsApp to ~240 eligible students. Sixty-four volunteers consented and were randomized by an independent researcher into two strata (3rd and 4th year), then assigned to:

Experimental group (n=32)

Control group (n=32) Participant confidentiality was maintained using four-digit codes to pair pre-/post-tests.

Intervention (Experimental Group)

A three-session structured education program on infant massage delivered by an experienced instructor holding certifications in breastfeeding counseling (200 h) and PIOMI. Sessions lasted 30-45 minutes each with 15-20-minute breaks and included:

Orientation and Pre-test: study overview, consent, completion of baseline forms.

Education Session: content prepared from current literature and adult-learning principles; video demonstration covering massage stages (preparation, technique, safety, communication).

Supervised Practice and Post-test: guided practice on a mannequin with feedback; completion of post-test.

Practical skills were observed with a simple checklist to ensure correct sequence and safety (no scoring is reported as an outcome).

Comparator (Control Group) No infant-massage training during the study period. Control participants completed the same baseline and post-test knowledge assessments over the same timeframe.

Outcomes and Measures

Primary Outcome: Infant Massage Knowledge score, measured at baseline and immediately post-intervention using the 15-item Baby Massage Knowledge Form (yes/no format) with three subdomains:

Preparation before massage (5 items)

During-massage practices (6 items)

Post-massage practices (4 items) Higher total scores indicate greater knowledge.

Data Collection and Management Forms were administered in paper or secure digital format and linked using participant codes. Data were checked for completeness before entry. Only the research team had access to the de-identified dataset.

Statistical Analysis Analyses were performed in SPSS v26. Descriptive statistics summarized demographics (means, SDs, frequencies). Group equivalence at baseline was examined with chi-square tests for categorical variables and appropriate parametric/non-parametric tests for continuous variables. The primary analysis compared post-test knowledge between groups (independent samples t-test or non-parametric equivalent as required). Within-group pre/post change was assessed with paired t-tests (or non-parametric equivalent). Two-sided α = 0.05 defined statistical significance.

Results (as completed study) Groups were comparable at baseline in age, income level, residence type, family type, prior awareness of infant massage, and information sources. Pre-test scores did not differ significantly between groups. Post-test scores were significantly higher in the experimental group than the control group, and the experimental group showed a significant pre/post increase; the control group showed only a small, non-significant change. These findings support the effectiveness of the brief structured training in improving infant-massage knowledge among midwifery students.

Ethical Considerations Ethics approval was obtained from the Atatürk University Non-Interventional Clinical Research Ethics Committee (Approval No. B.30.2.ATA.0.01.00/45, Date: 07 June 2024). Participation was voluntary, and written or verbal informed consent was obtained. The study involved minimal risk and confidentiality was maintained through coded data. No Data Monitoring Committee was required due to the short duration and low-risk nature of the study.

Data Monitoring and Harms No investigational drugs or devices were used. No adverse events were expected or observed. Any concerns raised by participants would have been documented and reported to the ethics committee per institutional policy.

Protocol Deviations None affecting primary outcome collection or analysis were recorded.

Dissemination Aggregate results will be shared through academic publications and presentations. No individual participant data are planned for public sharing.

Significance and Implications A short, structured classroom program combining video demonstration and supervised mannequin practice produced a meaningful gain in knowledge. Incorporating such modules into midwifery curricula may strengthen neonatal care competencies and support consistent, safe parent education on infant massage.

Limitations Single-institution sample may limit generalizability; outcomes focused on knowledge rather than long-term skill retention or clinical behaviors; immediate post-test timing prevents conclusions about durability of learning. Future studies should include multi-site cohorts, longer follow-up, and observational assessments of skills in clinical settings.

Current Study Status Enrollment and data collection are complete; analyses are finalized. Overall recruitment status: Completed. Study start: April 2024 (Actual). Primary completion: May 2024 (Actual). Study completion: June 2024 (Actual).

ELIGIBILITY:
Inclusion Criteria:

* Midwifery students enrolled in the 3rd or 4th year of study.
* Completed coursework in Child Health and Diseases Nursing and Neonatal Health.
* Literate in Turkish.
* Voluntarily agreed to participate and provided written and/or verbal informed consent.

Exclusion Criteria:

* Withdrew participation before completing data collection.
* Missing pre-test or post-test data.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-06-09 (Actual)

PRIMARY OUTCOMES:
Infant Massage Knowledge Score | Measured before training (pre-test) and after training (post-test, immediately after intervention)
  Change in participants' knowledge about infant massage before and after the educational intervention. Knowledge is assessed using the Infant Massage Knowledge Questionnaire (Gürol, 2010), which includes 15 yes/no items divided into three subscales: preparation, application, and post-application phases.

SECONDARY OUTCOMES:
Knowledge Retention Score | 1 month after the intervention (if follow-up conducted).
  Retention of infant massage knowledge measured at follow-up (if applicable) using the same Infant Massage Knowledge Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Faculty of Health Sciences, Department of Midwifery, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study involved educational interventions among students and collected only anonymized group data. No individual participant data (IPD) will be shared.